CLINICAL TRIAL: NCT00769964
Title: A First in Human Study Consisting of a Two-Part, Double-Blind, Placebo-Controlled, Escalating Single and Multiple Dose Study of VA111913 TS in Adult Non-Pregnant Women Volunteers With a Single Dose, Open, Fed vs. Fasting Crossover Phase
Brief Title: VA111913 TS: First in Human Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vantia Ltd (Industry)
Responsible Party: Acting Medical Director, Charles River Clinical Services
Purpose: Treatment
Other Study IDs: 913-001
Record Dates: First submitted 2008-10-08; First posted 2008-10-09 (Estimated); Last update posted 2009-06-25 (Estimated); Status verified 2009-06

CONDITIONS: Dysmenorrhea
Keywords: Healthy (Dysmenorrhea)
MeSH Terms: conditions — Dysmenorrhea

INTERVENTIONS:
Drug: VA111913 TS / placebo

SUMMARY:
This is a first-in-human study of VA111913 TS, a new chemical entity being developed for the treatment of dysmenorrhea. This study is designed to investigate determine the safety, tolerability and pharmacokinetics of VA111913 TS after single and multiple doses in healthy non-pregnant female volunteers of child bearing age.

DETAILED DESCRIPTION:
VA111913 TS is a selective V1a-receptor antagonist. The hypothesised mechanism of action of a V1a receptor antagonist in dysmenorrhea has been described in literature. Contractions of the uterine muscle are required for normal menstruation. Women with dysmenorrhea have increased uterine myometrial tone and contractions and decreased blood flow to the uterus. These abnormalities have been shown to lead to the pain experienced in dysmenorrhea. Thus, if a drug is able to reduce the hyperreactivity of the uterus to physiological levels then the pain experienced in dysmenorrhea may be controlled. In humans, vasopressin, via the V1a receptor, is able to potently induce contractions in both uterine smooth muscle and uterine blood vessels. Thus, a V1a receptor antagonist will potentially inhibit these contractions and in turn reduce the pain experienced in dysmenorrhea.

ELIGIBILITY:
Inclusion Criteria:

* Healthy females 18 to 45 years of age.
* Subjects must have a negative pregnancy test at screening and admission. Using acceptable form of contraceptive during and after study.

Exclusion Criteria:

* Administration of any IMP within 12 weeks before entry to the study or any prescribed medicine within 14days of the study.
* Any clinically important medical disease, condition or abnormal laboratory test results.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 98 (Actual)
Dates: Start 2008-09; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Charles River Clinical Services, Edinburgh, United Kingdom